CLINICAL TRIAL: NCT05094804
Title: A Phase 1-2 Study of OR2805, a Monoclonal Antibody Targeting CD163, Alone and in Combination With Anticancer Agents in Subjects With Advanced Malignancies
Brief Title: A Study of OR2805, a Monoclonal Antibody Targeting CD163, Alone and in Combination With Anticancer Agents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OncoResponse, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR2805-101
Record Dates: First submitted 2021-09-27; First posted 2021-10-26 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Tumor, Solid; Malignant Neoplasm; Metastatic Cancer; Advanced Solid Tumor; Non Small Cell Lung Cancer; Melanoma; Head and Neck Squamous Cell Carcinoma; Leiomyosarcoma; Liposarcoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Leiomyosarcoma; Liposarcoma | interventions — cemiplimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OR2805 monotherapy and combination therapy dose-escalation phase (Part A) (Experimental): Escalating repeated doses of OR2805 by IV administration as monotherapy or in combination with cemiplimab or docetaxel in subjects with advanced solid tumors. OR2805 will be administered once every 3 weeks (Q3W) or once-weekly (QW) for 3 weeks as an IV infusion over 30 minutes.
  Cemiplimab will be administered as an IV infusion at a dose of 350 mg.
  Docetaxel will be administered as an IV infusion at a dose of 75 mg/m2.
  Interventions: Drug: OR2805; Drug: Cemiplimab; Drug: Docetaxel
- OR2805 monotherapy and combination therapy dose-expansion phase (Part B) (Experimental): OR2805 administered IV at the RP2D and dosing regimen identified in Part A as monotherapy or in combination with cemiplimab or docetaxel in subjects with NSCLC and melanoma.
  Cemiplimab will be administered as an IV infusion at a dose of 350 mg.
  Docetaxel will be administered as an IV infusion at a dose of 75 mg/m2.
  Interventions: Drug: OR2805; Drug: Cemiplimab; Drug: Docetaxel
- OR2805 biological effects phase (Part C) (Experimental): OR2805 administered IV at the RP2D and dosing regimen identified in Part A as monotherapy to determine the mechanism of action and potential predictors of response and pharmacodynamic markers in subjects with liposarcoma, leiomyosarcoma, or SCCHN or are not otherwise eligible for Cohort B.
  Interventions: Drug: OR2805

INTERVENTIONS:
Drug: OR2805 — IgG1 monoclonal antibody that binds specifically to the CD163 protein.
Drug: Cemiplimab — IgG4 mAb that binds to PD-1 and blocks its interaction with PD-L1 and PD-L2.
  Other Names: Libtayo
  Arms: OR2805 monotherapy and combination therapy dose-escalation phase (Part A); OR2805 monotherapy and combination therapy dose-expansion phase (Part B)
Drug: Docetaxel — An antineoplastic agent that acts by disrupting the microtubular network in cells that is essential for mitotic and interphase cellular functions.
  Other Names: Taxotere
  Arms: OR2805 monotherapy and combination therapy dose-escalation phase (Part A); OR2805 monotherapy and combination therapy dose-expansion phase (Part B)

SUMMARY:
This is an open-label, multicenter, first-in-human dose-escalation and expansion Phase 1-2 study designed to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of OR2805 administered as a monotherapy and in combination with anti-cancer agents in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This Phase 1-2 study is designed to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of OR2805, a fully human IgG1 antibody that binds specifically to CD163, in subjects with advanced solid tumors. The study consists of three parts:

* Part A: a dose-escalation phase to determine the maximum-tolerated dose (MTD), maximum achievable dose, or recommended phase 2 dose (RP2D) of OR2805 given alone or in combination with cemiplimab or docetaxel in a maximum of approximately 54 subjects.
* Part B: an expansion phase in subjects with melanoma or non-small cell lung cancer (NSCLC) treated with OR2805 as monotherapy at the RP2D or OR2805 in combination with cemiplimab or docetaxel. Up to approximately 20 subjects will be treated in each arm of the 3 Part B cohorts to further characterize safety and determine the preliminary anti-tumor activity.
* Part C: a biology cohort of up to approximately 40 subjects at the RP2D to determine the mechanism of action and potential predictors of response and pharmacodynamic markers in subjects with liposarcoma, leiomyocarcoma, or squamous cell carcinoma of the head and neck (SCCHN) or are not otherwise eligible for Part B. All subjects in Part C will undergo biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the subject prior to conducting study-specific procedures.
2. Male or female subjects ≥ 18 and ≤ 100 years of age.
3. Histological diagnosis as follows:

   1. Part A (dose-escalation Cohorts A1-A3): histological diagnosis of any type of carcinoma, sarcoma, or melanoma with progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy.
   2. Part B (expansion Cohorts B1-B3): histological diagnosis of the relevant tumor type (NSCLC or melanoma) with advanced/metastatic disease not amenable to local therapy.

   a. Part C (biology cohort): histological or cytological diagnosis of any type of carcinoma, sarcoma, or melanoma with progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy. At least 10 subjects each must have a diagnosis of SCCHN, dedifferentiated liposarcoma, or leiomyosarcoma with prior treatment described below.
4. Prior therapies:

   a. Part A (dose-escalation) i. Subjects must have experienced PD on an established standard systemic anti-cancer therapy for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds. Subjects must have no available proven curative or life-prolonging therapies.

   b. Part B (dose-expansion) i. Part B1 subjects (NSCLC) must have received platinum-based therapy, unless contraindicated, and a PD-1 or PD-L1 inhibitor. Subjects eligible for targeted therapies to EGFR, ALK, ROS, RET or NTRK (e.g., crizotinib) must have previously received and exhausted such therapies. Prior therapies may have been administered alone or in combination. Subjects must have received prior PD-(L)1-based therapy as the most recent prior therapy and demonstrated progression while on that therapy.

   ii. Part B2 subjects (NSCLC) must have received platinum-based therapy and a PD-1 or PD-L1 inhibitor unless contraindicated. Subjects eligible targeted therapies to EGFR, ALK, ROS, RET or NTRK (e.g., crizotinib) must have exhausted such therapies. Prior therapies may have been administered alone or in combination. Part B2 subjects may have received a total of 3 lines of prior therapy and are not required to have received a PD-(L)1-based therapy as the most recent therapy.

   iii. For melanoma: subjects must have received a PD-1 inhibitor, alone or in combination with another immunotherapy. Eligible subjects may have received BRAF- and MEK-targeted therapies. Subjects must have received prior PD-1-based therapy as the most recent therapy and demonstrated radiographic progression while on that therapy.

   c. Part C (biology cohort): subjects other than those with liposarcoma, leiomyosarcoma, or SCCHN must have experienced PD on an established standard medical anti-cancer therapy for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds and must have no available demonstrated curative or life-prolonging therapies. Subjects with liposarcoma must have dedifferentiated liposarcoma, have received at least 1 prior systemic therapy, and require additional treatment. For leiomyosarcoma, subjects must have received at least 1 prior therapy for advanced or metastatic disease. For SCCHN, subjects must have received 1 prior line of chemotherapy and a PD-1- or PD-L1-targeted agent alone or in combination with chemotherapy unless contraindicated. No more than 2 chemotherapy regimens in the advanced setting for SCCHN are allowed. All subjects must have demonstrated progression on the most recent line of therapy.
5. Subjects must have measurable disease per RECIST v1.1. Subjects in Part C must have at least one 1 lesion amenable to biopsy and that is not to be used for response assessment per RECIST v1.1.
6. If not postmenopausal or surgically sterile, subjects must be willing to practice at least one of the following highly effective methods of birth control for at least a menstrual cycle (or partner's menstrual cycle, for male subjects) before and for 3 months after study medication administration: (1) true abstinence, when this is in line with the preferred and usual lifestyle of the subject, from sexual intercourse with a member of the opposite sex; (2) sexual intercourse with vasectomized male/sterilized female partner; (3) hormonal female contraceptive (oral, parenteral, intravaginal, implantable, or transdermal) for at least 3 consecutive months prior to investigational product administration (when not clinically contraindicated as in breast, ovarian, and endometrial cancers); (4) use of an intrauterine contraceptive device or intrauterine hormone-releasing system.
7. Resolution of prior-therapy-related AEs (excluding alopecia and grade ≤ 2 peripheral neuropathy) to ≤ grade 1 per CTCAE v5.0, and no treatment for these AEs for at least 2 weeks prior to the time of enrollment. Electrolyte and hormonal supplementation may be used to treat these AEs provided the subject is stable on these supplements.
8. Minimum of 2 weeks since the last dose of other hormone therapy and 3 weeks since the last dose of other systemic cancer therapy or radiotherapy (> 4 weeks in case of nitrosoureas or radio-immuno conjugate therapy). Adjuvant hormonal therapy (for example tamoxifen) is allowed provided the original tumor diagnosis was more than 3 years before the first dose of study medication.
9. Subjects must have adequate organ function.
10. All subjects must be able to supply an archival tumor biopsy specimen. For Part C (biology cohort), subjects must consent to a newly obtained tumor biopsy (that can be biopsied based on Investigator's assessment) and to providing the acquired tissue for biomarker analysis. An additional on-treatment biopsy is required for subjects in Part C.
11. Subject is able and willing to comply with the protocol and the restrictions and assessments therein.

Exclusion Criteria:

1. Subject previously had a severe hypersensitivity reaction to treatment with another mAb.
2. Subject has ECOG PS > 2.
3. Life expectancy <12 weeks.
4. Prior organ or stem cell transplant.
5. Subjects with symptomatic ascites or pleural effusion.
6. Subject has a known active CNS primary tumor or metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no radiological evidence of new or enlarging brain metastases, and are off steroids or on a stable dose up to an equivalent of prednisone 10 mg/day for at least 15 days prior to first dose of study medication. Subjects who have symptoms consistent with CNS metastasis, must have a negative MRI during in the screening period.
7. Subject has a known history of a hematologic malignancy, malignant primary brain tumor, or another malignant primary solid tumor (other than that under study), unless the subject has undergone potentially curative therapy with no evidence of that disease for at least 3 years.
8. Recent or ongoing serious infection including the following:

   1. Any uncontrolled grade 3 or higher (per CTCAE v5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of OR2805. Routine antimicrobial prophylaxis is allowed.
   2. Uncontrolled infection with HIV. Subjects on stable HARRT therapy with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
   3. Known to be positive for hepatitis B surface antigen, or any other positive test for hepatitis B indicating acute or chronic infection. Subjects who are or have received anti-HBV therapy and have undetectable HBV DNA for at least 6 months prior to study entry are eligible.
   4. Known active hepatitis C as determined by positive serology and confirmed by PCR. Subjects on or having received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry.
   5. Known active or latent tuberculosis (testing at screening is not required).
9. Autoimmune disease or inflammatory condition requiring systemic therapy with exceptions as noted in exclusion criterion 10.
10. Use of systemic corticosteroids within 15 days or other immunosuppressive drugs within 30 days prior to start of the study, with the exception of corticosteroids as replacement therapy up to an equivalent of prednisone 10 mg/day which are allowed. Pretreatment with dexamethasone is allowed for subjects receiving OR2805 in combination with docetaxel. Inhaled, topical, or intraarticular steroids are allowed.
11. Subject has received an investigational product or been treated with an investigational device within 30 days prior to first administration of study medication.
12. For Part B:

    1. Known contraindication to receiving cemiplimab.
    2. Interstitial lung disease.
    3. Prior pneumonitis requiring systemic corticosteroid therapy.
    4. Receiving immunosuppressive therapy, with exceptions as noted in exclusion criterion 10.
    5. A history of severe immune-related adverse reactions from treatment with ipilimumab, defined as any grade 4 toxicity or grade 3 toxicity requiring corticosteroid treatment (> 10 mg/day prednisone or equivalent) for more than 12 weeks.
13. Concurrent therapy with anti-cancer or anti-neoplastic drugs, with the exception of adjuvant hormonal therapy, which is allowed provided the subject has undergone potentially curative therapy with no evidence of disease for at least 3 years.
14. History or clinical evidence of any surgical or medical condition that the Investigator judges as likely to interfere with the results of the study or pose an additional risk in participating, e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, autoimmune or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
15. Subjects who, at the time of signing informed consent, had a recent history (within the last year) of chronic substance abuse.
16. Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Safety and Tolerability | Screening to 90 days from last dose.
  The nature, frequency, and severity of adverse events and serious adverse events, treatment discontinuations due to toxicity, and clinical laboratory abnormalities; recording of infusion-related reactions; physical examination and ECG findings; vital sign measurements; ECOG performance status scores; markers of inflammation and immunogenicity.
Recommended Dose and Regimen (mono and combination therapy) | Screening to 90 days from last dose.
  Determination of the MTD or maximum achievable dose, and the RP2D.

SECONDARY OUTCOMES:
Pharmacokinetics of OR2805 | Day 1 of dosing through 21 days post last dose.
  Peak plasma concentration (Cmax).
Pharmacokinetics of OR2805 | Day 1 of dosing through 21 days post last dose.
  Area under the plasma concentration versus time curve (AUC).
Objective Response Rate (ORR) | Day 1 of dosing through every 90 after the last dose.
  ORR according to RECIST v1.1.
Disease Control Rate (DCR) | Day 1 of dosing through every 90 after the last dose.
  The percentage of subjects with a complete response, partial response, or stable disease for at least 2 consecutive tumor assessments.
Progression Free Survival (PFS) | Day 1 of dosing through every 90 after the last dose.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for PD or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - NEXT Austin, Austin, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No